CLINICAL TRIAL: NCT01178255
Title: Homeopathy for Depression: a Randomized, Partially Double-blind, Placebo Controlled, Four Armed Study DEP-HOM
Brief Title: Efficacy and Safety of Homeopathy for Moderate Depression (Acute Phase)
Acronym: DEP-HOM
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: recruitment difficulties
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Claudia M. Witt, Prof. Dr. med., Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DEP-HOM10; 2009-017458-11 (EudraCT Number)
Record Dates: First submitted 2010-08-09; First posted 2010-08-10 (Estimated); Last update posted 2012-07-10 (Estimated); Status verified 2012-07

CONDITIONS: Major Depression
Keywords: depression; homoeopathy
MeSH Terms: conditions — Depressive Disorder, Major; Depression

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Group 1 (Experimental)
  Interventions: Drug: homeopathic q-potencies; Other: homeopathic case history taking type I
- Group 2 (Experimental)
  Interventions: Drug: Placebo; Other: homeopathic case history taking type I
- Group 3 (Experimental)
  Interventions: Drug: homeopathic q-potencies; Other: homeopathic case history type II
- Group 4 (Experimental)
  Interventions: Drug: Placebo; Other: homeopathic case history type II

INTERVENTIONS:
Drug: homeopathic q-potencies — individualised homeopathic medicines
  Arms: Group 1; Group 3
Drug: Placebo — placebo
  Arms: Group 2; Group 4
Other: homeopathic case history taking type I — one special homeopathic technique for case history taking
  Arms: Group 1; Group 2
Other: homeopathic case history type II — another type of homeopathic case history taking
  Arms: Group 3; Group 4

SUMMARY:
To assess the two components of individualized homeopathic treatment for acute depression, i.e., to investigate the specific effect of individualized Q-potencies versus placebo and to investigate the effect of different approaches to the homeopathic case history taking(defined in this study as case history taking type I and II).

DETAILED DESCRIPTION:
Homeopathy is often sought by patients with depression. In classical homeopathy, the treatment consists of two main elements: the taking of the case history and the prescription of an individually selected homeopathic remedy. Homeopathic medicines are produced through sequential, agitated dilutions. A Q-Potency is prepared by grinding the raw material, followed by a process of consecutive 1:50.000 agitated dilutions.

Previous data suggest that individualized homeopathic Q-potencies were non inferior to the antidepressant fluoxetine in a sample of patients with moderate to severe major depression. The question remains whether individualized homeopathic Q-potencies have a specific therapeutical effect in acute depression as this has not yet been investigated.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of major depression by a psychiatrist,
* patients must not be currently taking antidepressants or anxiolytic drugs (with the exception of Lorazepam as rescue medication, maximal dose 1.5 mg/day)
* Capability and willingness to give informed consent and to comply with the study procedures will also be required

Exclusion Criteria:

* current mild episode of depression (HAM-D < 17)
* current severe episode of depression (HAM-D > 24)
* schizophrenia or other psychotic disorders
* bipolar affective disorder
* schizoaffective disorders
* alcohol or other substance abuse
* eating disorders
* a clinically significant (Diagnostic and Statistical Manual of Mental Disorders)-Axis II disorder
* severe depression, which previously motivated a suicide attempt
* a score of 4 or 5 in the Columbia-Suicide Severity Rating Scale (C-SSRS)up to three months before screening;
* a clinically significant acute or chronic disease that would hinder regular participation in the study
* treatment with antipsychotics, antidepressants, sedatives/hypnotics or mood stabilizers four weeks prior to the screening
* complementary or alternative treatment simultaneously to the study (for example, acupuncture, phytotherapy, etc.)
* homeopathic treatment eight weeks prior to study entry
* psychotherapy
* simultaneous participation in another clinical trial (the last participation in a previous clinical trial must be completed at least three months prior to screening)
* concomitant pregnancy or breastfeeding
* patients who are assumed to have a linguistic, intellectual or any other reason for not understanding the meaning of the clinical trial and for not complying with the necessary study procedures
* persons who have been institutionalized by a court order
* patients with an application for a pension

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2010-08; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
primary endpoint is the mean total depression score post treatment | six weeks
  total score on the 17-item Hamilton Depression Rating Scale - (HAM-D)

SECONDARY OUTCOMES:
mean total depression score during the treatment | two and four weeks
  total score on Hamilton Depression Rating Scale (HAM-D)
response and remission rates | two, four and six weeks
  response (decrease of 50% or more from baseline HAM-D score); remission (HAM-D scores ≤ 7)
Self-rated depression score | two, four and six weeks
  Beck Depression inventory (BDI) total score
quality of life assessment | two, four and six weeks
  total mean score on the SF-12 Health Survey
Safety | two, four and six weeks
  Adverse events will be collected during the study and will form part of the secondary endpoint data in determining the safety of homeopathic medicines. Adverse events and serious adverse events will be registered in accordance with the ICH-Guidelines for Good Clinical Practice

CONTACTS AND LOCATIONS:
Overall Officials: Claudia M. Witt, MD, Principal Investigator — Charite University, Berlin, Germany
Locations (1):
- Institute for Social Medicine, Epidemiology, and Health Economics, Charité University Medical Center Berlin, Germany, Berlin, State of Berlin, Germany

REFERENCES:
- [Background] Adler UC, Kruger S, Teut M, Ludtke R, Bartsch I, Schutzler L, Melcher F, Willich SN, Linde K, Witt CM. Homeopathy for depression--DEP-HOM: study protocol for a randomized, partially double-blind, placebo controlled, four armed study. Trials. 2011 Feb 14;12:43. doi: 10.1186/1745-6215-12-43. PMID 21320338
- [Derived] Adler UC, Kruger S, Teut M, Ludtke R, Schutzler L, Martins F, Willich SN, Linde K, Witt CM. Homeopathy for depression: a randomized, partially double-blind, placebo-controlled, four-armed study (DEP-HOM). PLoS One. 2013 Sep 23;8(9):e74537. doi: 10.1371/journal.pone.0074537. eCollection 2013. PMID 24086352